CLINICAL TRIAL: NCT06383676
Title: The Effect Of Functional Balance-Based Reaction Exercises On Improvement Of Physical Capacity And Cognitive Performance In Elderly Individual
Brief Title: Effect Of Functional Balance Exercise İn Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Fatma Kübra ÇEKOK, Asst.prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Older People; Exercise
Keywords: balance; reaction time; functional capacity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled study
Who Masked: Participant
Masking Description: Study participants are unaware of their assigned group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional balance based reaction exercise training. (Experimental): Functional balance-based balance reaction exercises will be integrated into functional balance exercises with the help of the BlazePod™ training device panel.
  Interventions: Other: Functional reaction balance training
- Functional balance training (Experimental): The exercises will consist of functional balance activities, such as maintaining a standing posture, transitioning from sitting to standing, walking and balancing on one leg.
  Interventions: Other: Functional balance training

INTERVENTIONS:
Other: Functional reaction balance training — The interventions will carried out two days a week and 40 minutes, for eight weeks.
  Arms: Functional balance based reaction exercise training.
Other: Functional balance training — The interventions will carried out two days a week and 40 minutes, for eight weeks.
  Arms: Functional balance training

SUMMARY:
The elderly population is increasing in Turkey and in the world. Many health problems, such as a decrease in physical and psychological abilities and an increase in chronic problems, occur with aging. It is important to encourage and support practices for the development of exercises to increase physical and cognitive capacity in order to early recognize and reduce the effects of problems that develop with aging. To the best of our knowledge, there is no exercise training to increase reaction time in the elderly in the literature.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. Volunteer participants over the age of 65 living in a nursing home in Ankara will be included in the study. The sample of the study will consist of 28 elderly individuals, as determined by power analysis. The participants will be randomly divided into two groups. One group (Group 1) will receive functional balance exercise training, and the other group (Group 2) will receive functional balance-based reaction exercise training. The participants socio-demographic information, cognitive level ( The Montreal Cognitive Assessment), executive function (Stroop Test), reaction time, physical performance (Four Step Square test, Short Physical Performance Battery, Time Up Go Test) and balance confidence (Falls Efficiency Scale) will be evaluated Evaluations will be repeated at baseline and 8 weeks later. The interventions will be carried out two days a week for 40 minutes for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 or above
* Minimum of 5 years of education
* Moca score of 21 or higher
* Capability to walk a minimum of 10 meters (with or without walking assistance if needed)

Exclusion Criteria:

* Moca test score 21 and below
* Having vision and hearing problems (which cannot be corrected with glasses or hearing aids)
* Having an orthopedic or neurological disease that prevents standing

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
The Montreal Cognitive Assessment (MoCA) | Eight weeks
  The Montreal Cognitive Assessment (MoCA) is a brief instrument developed for the screening of milder forms of cognitive impairment. A score is derived by summing the points from each successfully completed task, for a total range from 0 to 30 points; higher scores indicate better cognitive performance. The MoCA was developed to screen milder forms of cognitive impairment through the assessment of a wide range of cognitive functions, such as short-term memory, executive functions, visuospatial abilities, language, attention, concentration, working memory, and temporal and spatial orientation. It comprises a 1-page test, which requires a short administration time (10-15 minutes).
Stroop Test | Eight weeks
  The test consists of two cards, each containing 60 items, presented in six rows of 10 items. On the first card, there are small rectangles (0.5 x 1 cm) printed in red, green and blue. The second card contains names of the three colours (i.e., red, green and blue) printed in incongruent colours (e.g., the word 'red' is printed in blue ink). The Stroop test Çapa version consists of three parts: Stroop A, Stroop B and Stroop C. Stroop A. The first part of the test requires individuals to name the colours (i.e., red, green and blue) of the small rectangles as quickly as possible, following a sequence from left to right. If any sign of colour blindness or colour naming deficits is present, the test is discontinued. Stroop B. The second part of the test requires individuals to read as fast as possible the colour names (i.e., red, green, and blue) that are printed in incongruent ink colours.
  The Stroop test Çapa version consists of three parts: Stroop A, Stroop B and Stroop C. Stroop A. The
The Simple Reaction Time | Eight weeks
  The simple reaction time is measured using an electronic timing system (including a digital display, a light, and a button, and the protocol that has been described in the literature was followed . Each older is seated so that the resting arm was on the table in a quiet environment. The testing side's second index is placed 1 cm away from the button of the device. Then, the participants are asked to press the button when the visual or auditory input appeared. A total of 10 repetitions are recorded, and the mean score of the last 5 tests is further analyzed .. The visual and auditory reaction time is randomly assigned. The reaction time is recorded with 1/1,000 seconds of sensitivity.

SECONDARY OUTCOMES:
The Four Square Step Test (FSST) | Eight weeks
  The Four Square Step Test (FSST) has been widely used for evaluating dynamic balance in older populations. The FSST requires a stopwatch and four single-point sticks (SPS). Using the sticks resting flat on the floor to form a cross, the subject starts in one square, steps in one direction into each of the four squares, and then reverses direction back to the start.
The short physical performance battery (SPPB) | Eight weeks
  The short physical performance battery (SPPB) is a quick and useful tool for fall risk stratification among older primary care patients. The SPPB, a 3-part performance-based test (gait time, chair stand, and balance), was assessed at baseline. Each test is scored from 0 (inability to perform the task) to 4 points (best test performance) . The SPPB total score ranges from 0 (worst performance) to 12 points (best performance) and categorically evaluates performance in the tests using three or four classes of scores: three classes: 0-6 points (poor performance),
Timed Up and Go Test (TUG) | Eight weeks
  Timed Up and Go Test (TUG) has been recommended as a simple fall risk screening tool, primarily to identify people warranting more-detailed assessment of gait and balance. Measures the time taken (in seconds) for a person to rise from a chair with armrests, walk 3 meters with usual assistive devices, turn, return to the chair, and sit down
Falls Efficacy Scale ( FES) | Eight weeks
  Falls Efficacy Scale is widely used 16-item Falls Efficacy Scale (FES) evaluate the social dimension of fear of falling and refers almost exclusively to very basic activities of daily living, making it insensitive when used in active older persons. Each item is scored on a four-point scale: 1 = not at all concerned, 2 = somewhat concerned, 3 = fairly concerned and 4 = very concerned. A summary score is calculated by adding the score of each item, giving a scale ranging from 16 to 64 for the 16-item FES-I and from 7 to 28 for the seven-item FES-I. A low score indicates low fear of falling
Mini-BESTest: Balance Evaluation Systems Test | Eight weeks
  The Balance Evaluation Systems Test (BESTest) is a relatively new multi-task balance assessment developed to identify specific postural control problems (i.e., biomechanical constraints, stability limits, postural responses, anticipatory postural adjustments, sensory orientation, dynamic balance during gait, and cognitive effect). The Mini-BESTest is a 14-item performance-based measure of balance disorders.The total score ranged from 0 to 28, with higher scores denoting better balance ability.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Kübra ÇEKOK, Phd, Principal Investigator — Tarsus University
Locations (1):
- Fatma Kübra ÇEKOK, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No